CLINICAL TRIAL: NCT01124799
Title: Photosensitivity Trial. A Randomized, Double-blind, Double Dummy, Placebo- and Positive Controlled Phase I Trial to Evaluate the Photosensitizing Potential of TMC435 in Healthy Subjects.
Brief Title: TMC435-TiDP16-C125 - Study in Healthy Volunteers to Evaluate the Potential of TMC435 to Increase the Sensitivity of the Skin Towards Exposure to Sun Light
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tibotec Pharmaceuticals, Ireland (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR017158
Record Dates: First submitted 2010-05-13; First posted 2010-05-17 (Estimated); Last update posted 2013-05-06 (Estimated); Status verified 2013-05

CONDITIONS: Hepatitis C Virus
Keywords: Hepatitis C virus; TMC435-TiDP16-C125; TMC435-C125; TMC435; TMC435350; protease inhibitor; HCV; Hepatitis C; photosensitivity; phototoxicity
MeSH Terms: conditions — Hepatitis C; Photosensitivity Disorders; Dermatitis, Phototoxic | interventions — Simeprevir; Ciprofloxacin

ARMS (3):
- 001 (Experimental): TMC435 one morning TMC435 dose between 75 and 150 mg and a placebo dose at noon and in the evening for 9 days
  Interventions: Drug: TMC435
- 002 (Placebo Comparator): Placebo placebo dose in the morning at noon and in the evening for 9 days
  Interventions: Drug: Placebo
- 003 (Active Comparator): Ciprofloxacin one morning placebo dose and a noon and evening dose of ciprofloxacin 500 mg for 9 days
  Interventions: Drug: Ciprofloxacin

INTERVENTIONS:
Drug: TMC435 — one morning TMC435 dose between 75 and 150 mg and a placebo dose at noon and in the evening, for 9 days
  Arms: 001
Drug: Placebo — placebo dose in the morning, at noon and in the evening, for 9 days
  Arms: 002
Drug: Ciprofloxacin — one morning placebo dose and a noon and evening dose of ciprofloxacin 500 mg, for 9 days
  Arms: 003

SUMMARY:
The purpose of the study is to evaluate the potential effect of TMC435 on the sensitivity of the skin towards exposure to sunlight. TMC435 is a drug that is currently under development for treatment of chronic hepatitis C virus infection. This study will be conducted in healthy volunteers. Ciprofloxacin, a commonly used antibiotic, is used as a positive control as this drug is known to mildly increase skin sensitivity to exposure to sunlight. This study also evaluates the levels of TMC435 and ciprofloxacin in the blood circulation and the safety and tolerability of TMC435.

DETAILED DESCRIPTION:
This is a randomized (study drug assigned by chance), double blind (neither the study doctor, nor medical staff nor the healthy volunteer know the name of the assigned drug), double-dummy (all healthy volunteers take the same number of identically looking capsules, independent of the drug they have been assigned to), placebo- and positive-controlled (ciprofloxacin is a drug known to cause a mild photosensitive response) study. A total of 36 healthy volunteers will participate. Participants will be assigned to take TMC435 (one dose between 75 and 150 mg, once a day), TMC435-placebo (once a day) or ciprofloxacin (500 mg twice a day). The aim of this study is to look at the reaction of the skin after exposure to artificial sunlight when taking TMC435, ciprofloxacin or placebo. Study drug will be administered for 9 days. Phototesting (area of skin on your back will be exposed to artificial sunlight) will be conducted during 3 days before intake of study medication starts and during 3 days (Days 8, 9 and 10) during treatment. Skin reactions, general tolerability and safety of TMC435 will be assessed throughout the trial period (or longer if needed). Blood and urine samples will be taken at screening, on day 1, day 7, day 10 and at 2 follow-up visits. Blood levels of TMC435 and ciprofloxacin will be determined on Day 1, 5, 6, 7 (16 times), 8 (twice), 9 (twice) and 10. ECG and vital signs will be taken at screening, on day 1, twice on day 7, on day 10 and at 2 follow-up visits. A physical examination will be done at screening, on day 1, day 10 and at both follow-up visits. Volunteers assigned to the TMC435 group will receive a morning oral dose (dose between 75 and 150 mg) of TMC435 and a noon and evening oral dose of placebo, for 9 consecutive days. Volunteers assigned to the placebo group will receive oral placebo doses in the morning, at noon and in the evening, for 9 consecutive days. Volunteers assigned to the ciprofloxacin group will receive an oral morning placebo dose and a noon and evening oral dose of 500 mg ciprofloxacin, for 9 consecutive days.

ELIGIBILITY:
Inclusion Criteria:

* Skin type I to III
* No ultraviolet exposure on the back for 4 weeks prior to baseline phototesting
* Normal skin response during baseline phototesting
* Body Mass Index of 18.0 to 30.0 kg/m2
* Healthy based on a medical evaluation including medical history, physical examination, blood tests and electrocardiogram.

Exclusion Criteria:

* History of hypersensitivity to sunlight or artificial source of intense light, especially UV light
* history or currently active porphyria or lupus erythematosus
* Positive plasma porphyrin scan and lupus erythematosus antibodies
* Active skin disorders on the back where phototesting will be performed
* Infection with Hepatitis A, B or C virus
* Infection with the human immunodeficiency virus (HIV)
* Women who are pregnant or breastfeeding
* History of or any current medical condition which could impact the safety of the participant in the study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2010-07; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
The effect of TMC435 versus placebo on the sensitivity of the skin towards sun light | Final phototesting assessment will be done on day 9 and 10 during medication intake.

SECONDARY OUTCOMES:
Rate and extent of absorption of TMC435 and ciprofloxacin in the blood circulation | Determined on Day1, 5, 6, 7, 8, 9 and 10, with extensive pharmacokinetic testing on Day7.
Number of participants with Adverse Events as measures for Safety and Tolerability.. | Until last follow-up visit 30-35 days after last drug intake.
Number of Adverse Events (per type) as measures for Safety and Tolerability. | Until last follow-up visit 30-35 days after last drug intake.
Results of clinical laboratory evaluations as measures for Safety and Tolerability. | Until last follow-up visit 30-35 days after last drug intake.
Vital signs including ECG monitoring as measures for Safety and Tolerability. | Until last follow-up visit 30-35 days after last drug intake.

CONTACTS AND LOCATIONS:
Overall Officials: Tibotec Pharmaceuticals Clinical Trial, Study Director — Tibotec Pharmaceutical Limited